CLINICAL TRIAL: NCT06796634
Title: Effects of Cold Atmospheric Plasma (CAP) on Peritoneal Tumor Tissue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2024-0090; B6702024000142 (Other: University Hospital Ghent)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cold Atmospheric Plasma (CAP); J-Plasma; Peritoneal Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with peritoneal metastases undergoing surgery (CRS, debulking), irrespective of the origi (Experimental): * Surgery and application of CAP: at the start of surgery, an inventory is made of suitable tumor nodules that will be planned for resection. Nodules should have a maximal size of 2-3 mm, since it is unlikely that bigger lesions can be adequately treated with CAP.
  * Selected tumor nodules will be treated with the J-plasma device at the standard settings (Helium gas flow of 4 l/min, coagulation and cutting intensity at 35). The distance between the tip of the device and the tissue will be approx. 10 mm. Using a timer and footswitch, nodules will be treated at different power settings and durations:
    * 15 W, 30W, or 45W
    * 2, 5, or 10 seconds.
  * The treated nodules will be resected at least 30 minutes after plasma treatment, and the exact timing will be documented. The samples are split in half: one half is fixed in formalin for histology and immune histochemistry, and the other half is immediately processed for live/death staining using flow cytometry.
  Interventions: Device: J-plasma

INTERVENTIONS:
Device: J-plasma — * Surgery and application of CAP: at the start of surgery, an inventory is made of suitable tumor nodules that will be planned for resection. Nodules should have a maximal size of 2-3 mm, since it is unlikely that bigger lesions can be adequately treated with CAP.
  * Selected tumor nodules will be treated with the J-plasma device at the standard settings (Helium gas flow of 4 l/min, coagulation and cutting intensity at 35). The distance between the tip of the device and the tissue will be approx. 10 mm. Using a timer and footswitch, nodules will be treated at different power settings and durations:
    * 15 W, 30W, or 45W
    * 2, 5, or 10 seconds.
  * The treated nodules will be resected at least 30 minutes after plasma treatment, and the exact timing will be documented. The samples are split in half: one half is fixed in formalin for histology and immune histochemistry, and the other half is immediately processed for live/death staining using flow cytometry.

SUMMARY:
There are to date no studies available that have examined the effects of CAP on tumor tissue in patients. The aim of this study is to investigate these effects in patients undergoing surgery for peritoneal metastases. Tumor nodules will be treated with different durations and intensities of CAP before being surgically removed. The resected nodules will be analyzed for tumor vitality.

ELIGIBILITY:
Inclusion criteria:

* Patients with peritoneal metastases undergoing surgery (CRS, debulking), irrespective of the origin. Potential cancer types include ovarian cancer, colorectal cancer, and malignant peritoneal mesothelioma
* Written informed consent
* Age ≥ 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
- Histology: | 1 year
  Following resection, FFPE sections will be assessed morphologically, particularly for the extent of tumor necrosis using haematoxylin and eosin staining. IHC staining will be performed to investigate mechanisms of autophagia (p62 and LC3B), apoptosis (cleaved caspase 3) and proliferation (ki67).
  * Extent of tumor necrosis: morphological assessment
  * Proliferation: Ki67 via MIB1
  * Autophagia: p62 or LC3B
  * Apoptosis: Caspase 3 antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Ghent, Ghent, East-Flanders, Belgium